CLINICAL TRIAL: NCT05833373
Title: Transcutaneous Vagal Nerve Stimulation for the Treatment of Persistent Atrial Fibrillation (VAST-AF): a Randomized, Controlled, Blinded, Monocentric, Clinical Trial
Brief Title: Vagal Nerve Stimulation for the Treatment of Persistent AF
Acronym: VAST-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krankenhaus Hetzelstift (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Patrick Swojanowsky, Dr. med. Patrick Swojanowsky, Krankenhaus Hetzelstift
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Studie VAST-AF Swo
Record Dates: First submitted 2023-04-17; First posted 2023-04-27 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Vagal stimulation; Transcutaneous nerve stimulation; Autonomic nervous system; parasympathetic nervous system
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants are randomized 1:1 to either the verum- or the sham-group. Both device look similar and are used in the same way so the participants are blinded. This is achieved with a conducting and a non-conducting ear electrode.
  The care provider and the investigator is blinded as well. The researcher who randomises the patient is strictly separated from the investigator who is responsible for the follow-up. Only after the patient completed the last follow-up the outcome assessor will match the patient data with the affiliation to either the sham- or the verum-group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum group (Experimental): Verum group - active vagal stimulation with the stimulation device tVNS from tVNS Technologies GmbH. The stimulation is performed with an ear-electrode at the Tragus. Minimal stimulation duration is 1 hour per day for 3 months.
  Interventions: Device: Vagal stimulation with the device tVNS from tVNS Technologies GmbH
- Sham group (Sham Comparator): Sham group with ineffective vagal stimulation. Same stimulation procedure like in the verum group with the stimulation device tVNS from tVNS Technologies GmbH. The stimulation is performed with an ear-electrode at the Tragus, too. Minimal stimulation duration is 1 hour per day for 3 months, but with a non conducting ear electrode.
  Interventions: Device: Sham stimulation with the device tVNS from tVNS Technologies GmbH

INTERVENTIONS:
Device: Vagal stimulation with the device tVNS from tVNS Technologies GmbH — The tVNS device is used to stimulate the Ramus auricularis of the Nervus vagus with a dedicated ear electrode for at least one hour per day on a daily basis. Stimulation frequency is 20Hz, pulsewidth is 200µs and amplitude is determined individually.
  Arms: Verum group
Device: Sham stimulation with the device tVNS from tVNS Technologies GmbH — The tVNS device is used to stimulate the Ramus auricularis of the Nervus vagus with a dedicated ear electrode for at least one hour per day on a daily basis. In this case to perform a sham stimulation a non conducting ear electrode is used. The device is set to the same settings with a frequency of 20Hz, a pulsewidth of 200µs and an amplitude that is determined individually.
  Arms: Sham group

SUMMARY:
The goal of this clinical trial is to answer the question whether a transcutaneous stimulation of a certain nerve (Nervus vagus) with a dedicated device reduces the recurrence of the heart rhythm disorder atrial fibrillation.

Participants will receive a dedicated nerval stimulation device and will treat themselves on a daily basis for at least an hour per day. Treatment will last for 3 months. Researchers will compare this group with a similar group that uses an ineffective device. Both researcher and patients will be blinded so they do not know which device they will be using.

DETAILED DESCRIPTION:
This study is an investigator-initiated, monocentric, randomised, controlled and blinded trial. Patients with persistent atrial fibrillation and planned electrical cardioversion will be included. The participants are randomised to one of two groups - the verum-group or the sham-group. Both groups receive a dedicated stimulation device that stimulates transcutaneously the Ramus auricularis of the Nervus vagus at the area of the Tragus. The verum-group will receive an effective stimulation and the sham-group an ineffective one. The aim of this trial is to evaluate whether this stimulation could reduce the recurrence of atrial fibrillation or not. Therefore daily stimulation of at least one hour will be performed for overall three months. After that period the stimulation will be withdrawn and both groups will be compared. Then, after another three months without stimulation both groups will be compared again to evaluate if a potential effect of the initial stimulation persists.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation
* Planned electric cardioversion
* Sufficient oral anticoagulation for at least four weeks or
* Absence of thrombus in transoesophageal echocardiography
* Oral anticoagulation possible
* Able to sign informed consent
* Estimated life expectancy >1 year

Exclusion Criteria:

* Permanent atrial fibrillation
* Ablation therapy of supraventricular arrhythmias in the past
* Missing anticoagulation respective missing rule out of thrombus
* Inability to treat with oral anticoagulation
* Latent or manifest hyperthyroidism
* Acute infection with relevant clinical signs (temp > 38°C, significant elevated C-reactive protein or white blood cells)
* Inability to sign informed consent
* Preexisting pacemaker or implantable cardioverter defibrillator
* Recent vagal stimulation for other causes
* Recent intolerance of transcutaneous vagal stimulation
* Estimated life expectancy <1 year
* Acute coronary syndrome
* Haemodynamic instability
* Valvular atrial fibrillation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 6 months
  Defined as an episode of atrial fibrillation >30 seconds that is detected with ECG, holter-ECG or wearable (i.e. Apple Watch). ECGs are performed during follow-up visits or could be conducted by an other hospital or during an ambulatory medical contact.

SECONDARY OUTCOMES:
Reduction of symptoms due to atrial fibrillation | 6 months
  Assessed with the Atrial Fibrillation Severity Scale: AFSS V2
Significant alterations of parameters of the autonomous nervous system | 6 months
  Different parameters of the autonomous nervous system like heart rate variability and heart rate turbulence etc. are analyzed via ECG
Delay in recurrence of atrial fibrillation due to vagal stimulation | 6 months
  Comparison of the time interval to the first recurrence of atrial fibrillation between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Swojanowsky, MD, Principal Investigator — Krankenhaus Hetzelstift
Locations (1):
- Marienhaus Klinikum Hetzelstift, Neustadt, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No